CLINICAL TRIAL: NCT02230943
Title: American College of Rheumatology's Rheumatology Informatics System for Effectiveness
Brief Title: Rheumatology Informatics System for Effectiveness
Acronym: RISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American College of Rheumatology (Other)
Responsible Party: Sponsor
Other Study IDs: RISE
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Gout
Keywords: rheumatoid; arthritis; osteoarthritis; gout
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Gout; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The RISE Registry is an enhanced version of the ACR's Rheumatology Clinical Registry (RCR) and allows for a simplified entry process, while establishing a best-in-class resource to manage your patient population and improve patient care.

RISE provides participants with an infrastructure for robust quality improvement activities leading to improved patient outcomes, patient population management and quality reporting related to rheumatic diseases and drug safety. RISE gives physicians and researchers the information they need to optimize patient outcomes, meet reporting requirements, and make discoveries that advance rheumatology.

DETAILED DESCRIPTION:
RISE helps providers benchmark performances on key rheumatology clinical quality measures and align with best practice standards. The RISE benchmarking tool allows providers to view the details of their patient population against established rheumatology quality metrics. RISE allows access to aggregate data from other participating sites so providers can view their patient population in comparison to other RISE participants.

RISE is integrated into an electronic health records (EHR) system, bringing a single point of entry into one solution for filing for quality-based incentive payments, avoiding penalties, complying with reporting requirements and tracking caseloads for quality monitoring and improvement initiatives. RISE collects the data needed to meet current federal reporting requirements.

Participating in RISE helps push the field of rheumatology practice forward. RISE provides a source of information on patient outcomes and quality care for rheumatology leading to new discoveries, better understanding and a source of comparative effectiveness research.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older with one of the following diagnoses: rheumatoid arthritis, osteoarthritis, gout

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Controlling High Blood Pressure | one year
  Percentage of patients 18-85 years of age who had a diagnosis of hypertension and whose blood pressure was adequately controlled (<140/90mmHg) during the measurement period.

CONTACTS AND LOCATIONS:
Locations (1):
- American College of Rheumatology, Atlanta, Georgia, United States